CLINICAL TRIAL: NCT02389179
Title: Maintenance of Vitamin D Sufficiency With Oral Vitamin D Supplementation in Malaysian Women of Malay and Indian Ethnicity With Post Menopausal Osteoporosis
Brief Title: Determination of Vitamin D Dose to Maintain Sufficiency Amongst Indian and Malay Women in the Tropics
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sharifah Faradila bt Wan Muhamad Hatta (Other)
Collaborators: Universiti Teknologi Mara (Other)
Responsible Party: Sponsor-Investigator, Sharifah Faradila bt Wan Muhamad Hatta, Doctor, University of Malaya
Organization: University of Malaya (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Vitamin D
Record Dates: First submitted 2015-03-04; First posted 2015-03-17 (Estimated); Last update posted 2015-12-16 (Estimated); Status verified 2015-12

CONDITIONS: Vitamin D Deficiency
Keywords: Vitamin D Deficiency
MeSH Terms: conditions — Vitamin D Deficiency | interventions — Cholecalciferol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 25 000 IU monthly (Active Comparator): The dose stated above are doses of Vitamin D3/Cholecalciferol which is formulated as spray dried powder stabilized with DL-alpha tocopherol (dry vitamin D3 100 SD/S)(DSM Nutritional Products Switzerland Ltd). The spray dried powder will be diluted in 10 mls of water and ingested orally by subjects under direct supervision in a clinic setting.
  Interventions: Drug: Vitamin D3
- 50 000 IU monthly (Active Comparator): The dose stated above are doses of Vitamin D3/Cholecalciferol which is formulated as spray dried powder stabilized with DL-alpha tocopherol (dry vitamin D3 100 SD/S)(DSM Nutritional Products Switzerland Ltd).The spray dried powder will be diluted in 10 mls of water and ingested orally by subjects under direct supervision in a clinic setting.
  Interventions: Drug: Vitamin D3
- 50 000 IU bi-weekly (Active Comparator): The dose stated above are doses of Vitamin D3/Cholecalciferol which is formulated as spray dried powder stabilized with DL-alpha tocopherol (dry vitamin D3 100 SD/S)(DSM Nutritional Products Switzerland Ltd).The spray dried powder will be diluted in 10 mls of water and ingested orally by subjects under direct supervision in a clinic setting.
  Interventions: Drug: Vitamin D3

INTERVENTIONS:
Drug: Vitamin D3 — The drug/dosage of Vitamin D3 will be given monthly or bi-weekly depending on the type of arm that the subjects are randomised into under direct supervision.
  Other Names: Cholecalciferol

SUMMARY:
Much research on vitamin D status has focused on seasonal variations in serum 25(OH)D levels in populations living at high altitudes and those of light-skinned Caucasian extraction, with little work done in multi ethnic populations living closer to the equator with regards to Vitamin d supplementation, prevalence, predictors and associations of hypovitaminosis D - the assumption, perhaps being vitamin D deficiency is unlikely in locations of plentiful sunshine. There is a dearth of studies on Vitamin D status in a group of subjects at especially high risk of falls/fractures i.e. post-menopausal women with osteoporosis living in South-East Asia. It is possible that differences in geography and ethnicity/culture amongst women with post menopausal osteoporosis (PMO) in Malaysia may necessitate supplemental Vitamin D doses that differ from those prescribed to North American Caucasians.

There is no unified consensus on the dose of Vitamin D supplementation. Neither is there agreement on definitions of sufficiency with some researchers targeting levels of serum 25(OH)D of >20ng/ml and others aiming for levels above 30ng/ml. The Institute of Medicine (IOM) 2010 guidelines, aiming for a lower serum 25(OH)D target of 20ng/ml, advocates maintenance doses of 600 IU/day in Postmenopausal women aged 51-70 and 800 IU/day for those aged >70 years. On contrary, the Endocrine Society 2011 guidelines state that maintenance doses up to 1500-2000 IU/day may be required to attain a higher optimal target of >30ng/ml. On addition, the 2014 National Osteoporosis Foundation Guidelines recommended that the Vitamin D level should be brought up to approximately 30ng/ml, and to maintain at this level taking into account those with limited sun exposure, obese and dark skin individuals, the daily requirement ranges from 800-2000 IU/day.

The investigators therefore designed a prospective randomized controlled trial comparing efficacy and safety of a low (900 IU/day) and high (1800IU/day and 3300IU/day) maintenance dose of Cholecalciferol (Vitamin D3) amongst community dwelling Indian and Malay with PMO living in Kuala Lumpur, Malaysia.

Hypothesis of the study is despite abundant exposure to sunlight, which is the main Vitamin D supplier, those who dress conservatively and individuals with darker skin may require a higher dose of Vitamin D to maintain sufficiency (>30ng/ml).

DETAILED DESCRIPTION:
This randomized controlled trial will evaluate the appropriate dose of Vitamin D required to maintain Vitamin D sufficiency amongst Indian and Malay PMO women. The study will last for six months. 150 PMO women of Indian and Malay ethnicity will be randomly allocated into 3 different dosing regimens i.e. (a) 25 000 IU/monthly (≈900 IU/day), (b) 50 000 IU/monthly (≈1800 IU/day) and (c) 50 000 IU/fortnightly (≈3300 IU/day). Each group will be containing an equal amount of Indian and Malay Individuals. Subjects will be recruited from the osteoporosis clinic at UMMC.

Inclusion Criteria

1. Post menopausal Osteoporosis women receiving treatment from the Osteoporosis Clinic, University of Malaya Medical Centre, Kuala Lumpur.
2. Resident in Malaysia, of South Indian descent or Muslim Malay wearing headscarf
3. Baseline serum 25(OH)D levels > 20 ng/ml or 50 nmol/L

Exclusion Criteria

1. Secondary osteoporosis e.g. glucocorticoid induced osteoporosis
2. Metabolic bone disease e.g. hypercalcaemia, primary hyperparathyroidism, hyperthyroidism, hypothyroidism, Paget's disease
3. Medications that interfere with bone / vitamin D metabolism e.g. hormone replacement therapy (HRT), Recombinant human parathyroid hormone i.e. Teriparatide, glucocorticoids, rifampicin and anticonvulsants
4. Calculated Creatinine Clearance of < 60 mls/min
5. Liver disease and Malabsorptive Diseases e.g. celiac disease, radiation, enteritis, active inflammatory bowel disease
6. Malignancy

All patients who fulfils the inclusion and exclusion criteria will be offered participation in the study and written consent will be obtained.

During the first visit blood samples will be taken and all relevant data will be obtained via an interview and questionnaire. Blood samples taken include total 25(OH)D, calcium, phosphate, albumin and PTH levels as well as full blood count, renal and liver function. Twenty-four hour urine calcium levels will also be measured.

A detailed past medical history and medication history focusing on use of bone-related therapies will be taken. Subjects will be requested to record medications that could affect vitamin D metabolism, e.g. glucocorticoids, Recombinant human parathyroid hormone i.e. Teriparatide, Hormone Replacement Therapy, Rifampicin and anticonvulsants. All calcium, vitamin D and multivitamin supplements taken within 3 months prior to the clinic visit will also be recorded.

Von Luschan scale will be used to determine the skin colour group that the patient belongs to. This scale contains 36 opaque glass tiles which is compared with the subject's skin on the back of the hands.

A validated sun exposure questionnaire evaluating amongst other things time spent outdoors with/without sun protection, body parts exposed to sun and travel in sunny areas; will be filled in with the help of a trained interviewer. Subsequently, the rule of nines will be used to calculate skin sun exposure. This number will be multiplied by the reported average sun exposure per week without sunscreen to calculate the sun exposure index. The subject's most recent dual x-ray absorptiometry results will be recorded.

All patients will receive advice on optimal sun exposure (10-20 minutes of sun exposure daily without sun block depending on gradations of skin colour) and dietary calcium requirements (1000 mg/day of elemental calcium) for treatment of osteoporosis.

A detailed diet history focusing on foods high in Vitamin D and calcium from a validated questionnaire will be obtained.

Subjects with 25(OH)D level of < 20ng/ml will initially receive a loading dose of 50 000 IU of Vitamin D3 weekly for 8 weeks as is standard clinical practice as recommended by the 2011 Endocrine Society guidelines, and serum 25(OH)D will be measured again after 8 weeks to ensure that levels are above 20ng/ml. They will then undergo an 8 weeks washout period in which the subjects will receive 25 000 IU of Vitamin D3 monthly for two months prior to randomization. If subjects are already > 20ng/ml at baseline they will proceed straight to randomisation.

All subjects will cease any previous over the counter Vitamin D supplements at study start. Thereafter subjects will be block randomized to either Vitamin D3 25 000 IU monthly, 50 000 IU monthly or 50 000 IU fortnightly of oral Cholecalciferol (Vitamin D3). Serum 25(OH)D, calcium, phosphate, iPTH and serum albumin will be measured again at 8, 16 and 24 weeks. At 24 weeks, 24 hour urine calcium will be measured again.

Any concomitant medications or adverse events will be recorded at every study visit at 4 weekly intervals.

All subjects will be assigned to receive 1g of calcium carbonate daily. Oral Cholecalciferol (powdered) will be ingested under direct supervision during study visits. Each dose of Cholecalciferol will be diluted in 10 mls of water. The Cholecalciferol used in this study is formulated as spray dried powder stabilized with DL-alpha tocopherol (dry vitamin D3 100 SD/S)(DSM Nutritional Products Switzerland Ltd).

ELIGIBILITY:
Inclusion Criteria:

1. Post menopausal osteoporosis woman receiving treatment from the Osteoporosis Clinic, University of Malaya Medical Centre, Kuala Lumpur.
2. Resident in Malaysia, of South Indian descent or Muslim Malay wearing headscarf
3. Baseline serum 25(OH)D levels > 20 ng/ml

Exclusion Criteria:

1. Secondary osteoporosis e.g. glucocorticoid induced osteoporosis
2. Metabolic bone disease e.g. hypercalcaemia, primary hyperparathyroidism, hyperthyroidism, hypothyroidism, Paget's disease
3. Medications that interfere with bone / vitamin D metabolism e.g. recombinant human parathyroid hormone i.e. Teriparatide, hormone replacement therapy (HRT), glucocorticoids, rifampicin and anticonvulsants
4. Calculated Creatinine Clearance of < 60 mls/min
5. Liver disease and Malabsorptive Diseases e.g. celiac disease, radiation, enteritis, active inflammatory bowel disease
6. Malignancy

Ages: 45 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2014-08; Primary Completion 2016-07 (Estimated); Study Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
Measuring optimal Vitamin D dose required to maintain vitamin D sufficiency (Serum 25(OH)D >30ng/ml in Malay and Indian PMO women. | 6 months
  This Randomised Control Trial will evaluate the appropriate dose of Vitamin D required to maintain sufficiency amongst Post Menopausal Malay and Indian descent Osteoporosis women.

CONTACTS AND LOCATIONS:
Overall Officials: Shireene Ratna Vethakkan, MBBS,MMED,MD, Principal Investigator — University of Malaya Medical Centre
Locations (1):
- University of Malaya Medical Centre, Kuala Lumpur, Kuala Lumpur, Malaysia